CLINICAL TRIAL: NCT00137306
Title: Translating Depression Guidelines Into Substance Abuse Treatment
Brief Title: Facilitating the Adoption of Evidence-Based Depression Management in Substance Use Treatment Programs
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: SUT 02-211
Record Dates: First submitted 2005-08-25; First posted 2005-08-29 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2007-02

CONDITIONS: Mood Disorders; Substance-Related Disorders
Keywords: Guideline Adherence; Quality Assurance, Health Care
MeSH Terms: conditions — Mood Disorders; Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Other)
  Interventions: Procedure: Facilitate evidence-based treatment for depression

INTERVENTIONS:
Procedure: Facilitate evidence-based treatment for depression

SUMMARY:
Comorbid depression has been consistently linked to worse outcomes for patients in substance abuse treatment programs. Practice guidelines recommend pharmacotherapy for comorbid depression if symptoms persist after a 4-week "wash-out" period for detoxification (e.g., Veterans Health Administration; American Psychiatric Association). Medications may be considered earlier if a patient has current symptoms and a history of major depressive disorder (MDD) during periods of sobriety. Current efficacy data suggest that antidepressant medication can improve both depression and substance use outcomes among comorbid patients Guideline-concordant use of antidepressant medication for persons with comorbid substance use and depressive disorders, however, is not routine in many VA substance abuse treatment settings.

DETAILED DESCRIPTION:
Background:

Comorbid depression has been consistently linked to worse outcomes for patients in substance abuse treatment programs. Practice guidelines recommend pharmacotherapy for comorbid depression if symptoms persist after a 4-week "wash-out" period for detoxification (e.g., Veterans Health Administration; American Psychiatric Association). Medications may be considered earlier if a patient has current symptoms and a history of major depressive disorder (MDD) during periods of sobriety. Current efficacy data suggest that antidepressant medication can improve both depression and substance use outcomes among comorbid patients Guideline-concordant use of antidepressant medication for persons with comorbid substance use and depressive disorders, however, is not routine in many VA substance abuse treatment settings.

Objectives:

This study seeks to develop, implement, and test an organizational intervention in VA substance abuse treatment settings to establish guideline-concordant treatment of comorbid depression. The intervention will assist "intervention" programs in their own implementation of a guidelines-based treatment algorithm to improve the recognition of depression and initiation of pharmacotherapy.

Methods:

Substance abuse treatment programs in the South Central VISN were matched on program characteristics and current depression management practices (n = 4), and "intervention" sites were randomly chosen from each pair. Phase 1 (now completed) of the study analyzed the barriers and facilitators to translation of depression management in participating facilities, and used these data to inform the development of the translation intervention, its implementation tools, and the depression algorithm. The translation intervention adopted in this plan was based on the PRECEDE model of organizational behavior change and included provider education, use of local champions, feedback of screening data, and patient education/activation. The depression management algorithm and intervention was developed with input from programs staff and an Advisory Panel of depression management and translation experts. Phase 2 of the study implemented and tested the intervention. The evaluation in examining program- and provider-level outcomes. Program-level outcomes include feasibility, extent of adoption of the algorithm, and provider/organizational attitudes and beliefs about the intervention's design and effectiveness. Patient-level outcomes include depressive symptoms, substance use outcomes, medication adherence, quality of life, and services use.

Status:

Phase 1 of the study is complete. Phase 2 is near complete.

ELIGIBILITY:
Inclusion Criteria:

Programs: VA's offering residential or intensive outpatient treatment for substance-related disorders in VISN 16 Patients: Veterans in residential or intensive outpatient treatment for substance-related disorders; positive screen for non-substance-induced depressive disorder

Exclusion Criteria:

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2004-01; Primary Completion 2006-10 (Actual); Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
Program: extent, quality of adoption of protocolPatient: scores on-depression, substance use, and functioning scales

SECONDARY OUTCOMES:
Programs: Staff satisfaction with protocol/intervention Patients: medication adherence

CONTACTS AND LOCATIONS:
Overall Officials: Geoffrey M. Curran, PhD, Principal Investigator — Central Arkansas Veterans Healthcare System Eugene J. Towbin Healthcare Center, Little Rock, AR
Locations (5):
- United States (5):
  - Central Arkansas Veterans Healthcare System Eugene J. Towbin Healthcare Center, Little Rock, AR, No. Little Rock, Arkansas
  - Southeast Louisiana Veterans Health Care System, New Orleans, LA, New Orleans, Louisiana
  - VA Gulf Coast Veterans Health Care System, Biloxi, Mississippi
  - G.V. (Sonny) Montgomery VA Medical Center, Jackson, MS, Jackson, Mississippi
  - Oklahoma City, OK, Oklahoma City, Oklahoma

REFERENCES:
- [Result] Curran GM, Mukherjee S, Allee E, Owen RR. A process for developing an implementation intervention: QUERI Series. Implement Sci. 2008 Mar 19;3:17. doi: 10.1186/1748-5908-3-17. PMID 18353186
- [Result] Curran GM, Kirchner JE, Worley M, Rookey C, Booth BM. Depressive symptomatology and early attrition from intensive outpatient substance use treatment. J Behav Health Serv Res. 2002 May;29(2):138-43. doi: 10.1007/BF02287700. PMID 12032971